CLINICAL TRIAL: NCT05928364
Title: Buccal Mucosal Graft for Onlay Ureteroplasty in the Management of Proximal Ureteral Stricture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Buccal graft ureteroplasty
Record Dates: First submitted 2023-05-22; First posted 2023-07-03 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Stricture Ureter
Keywords: Buccal mucosa; Stricture; ureteroplasty
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Patients with inclusion criteria of uretral stricture will be treated with open uretroplasty with buccal graft and omental wrapping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Buccal mucosa graft for ureteral stricture (Experimental): Patients with inclusion criteria of ureteral stricture will be treated with open ureteroplasty with buccal graft and omental wrapping.
  Interventions: Procedure: Buccal mucosa for proximal ureter stricture

INTERVENTIONS:
Procedure: Buccal mucosa for proximal ureter stricture — Patients with inclusion criteria of uretral stricture will be treated with open uretroplasty with buccal graft and omental wrapping

SUMMARY:
Onlay uretroplasty with either grafts or flaps has been attempted by many reconstructive urologists, ln particular buccal mucosa graft (BMG) ureteroplasty has been reported by many centers and has shown its feasibility and safety

DETAILED DESCRIPTION:
In cases of long segment upper ureteral stricture, more advanced surgical techniques, such as renal mobilization and downward nephropexy, ileal ureter replacement, transureteroureterostomy, and autotransplantation of the kidney, are necessary to provide a tension-free anastomosis.

Autotransplantation of the kidney needs more efforts, more experts and may lead to significant renovascular complications.

Also, there is severe metabolic and intestinal complications are associated with using of long intestinal segment in the management of ureteral stricture [9].

These previous side effects and difficulties make the management of long upper and middle ureteral strictures more complicated and indicate other lines of management urgently.

Even the ureteral stricture still not patent enough to drain urine but still, we can use it as a ureteral plate with little affection of its vascularity. Based on this theory an onlay repair technique was emerged.

Onlay uretroplasty with either grafts or flaps has been attempted by many reconstructive urologists, ln particular buccal mucosa graft (BMG) ureteroplasty has been reported by many centers and has shown its feasibility and safety.

ELIGIBILITY:
Inclusion Criteria:

* Proximal ureteral stricture or uretropelvic junction obstruction (UPJO) which are not amenable for primery anastmosis.

Exclusion Criteria:

* Buccal graft contraindications as i. Active oral infections ii.Oral cancers like cancers of lips, tongue or cheeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-11 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Restoration of ureteric patency. | 6 months post-operative
  Restoration of ureteric patency as assessed by contrast study (intravenous urography) and ureteroscope.

SECONDARY OUTCOMES:
Pain relief after surgery | 6 months post-operative
  Relief of pain measured by Visual Analog Score for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided